CLINICAL TRIAL: NCT02162199
Title: A Phase 1, Double-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Escalating Oral Doses of Debio 1450 in Healthy Subjects
Brief Title: A Single Dose Study of Debio 1450 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Debio 1450-102; 217596 (Other: CRO)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Bacterial Infections
Keywords: Antibiotic; Antibiotic Resistant Bacterial Infection
MeSH Terms: conditions — Bacterial Infections | interventions — afabicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Debio 1450 (Experimental): Debio 1450 40 mg, capsules, orally, once in the morning under fasted conditions
  Interventions: Drug: Debio 1450
- Placebo (Placebo Comparator): Placebo 0 mg, matching capsules, orally, once in the morning under fasted conditions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Debio 1450 — Single sentinel dosing of 40 mg per unit capsules is planned to escalate from 80 mg to 160, 320, 480, 640 and 800 mg, per respective dosing group. Doses may be modified based on review of available safety and pharmacokinetic (PK) data.
  Arms: Debio 1450
Drug: Placebo — Matching single sentinel dosing of placebo capsules is planned to escalate from 2 capsules to 4, 8, 12, 16 and 20 capsules, per respective dosing group. The number of capsules will match those delivering Debio 1450 for the group, as those doses may be modified based on review of available safety and pharmacokinetic (PK) data.
  Arms: Placebo

SUMMARY:
The sponsor is trying to develop a medicine for infections that are not cured by regular antibiotics. They have an experimental drug called Debio 1450 that may work. They need about 48 healthy adults to volunteer for this study.

This study looks at what the body does to the drug. It measures how the amount of drug in blood and urine changes over time.

From the screening visit through the follow-up visit may be up to 40 days. Volunteers go to the clinic in Baltimore for a screening visit. The study doctor chooses qualified volunteers to participate or serve as alternates. Alternates might not actually complete the study procedures.

The study doctor divides participants into groups of eight. Six receive Debio 1450 and 2 receive Placebo. The drug each participant receives is decided by chance - like flipping a coin.

Eligible volunteers check into the clinic for testing and those chosen to participate remain for a 5-day/ 4-night stay. The clinic serves standard meals, except when fasting is required. Participants must stay at the clinic for the length of the study.

This study is a "dose escalation" study. That means that if no safety concerns come up a new group starts. Each new group of eight participants receives more capsules.

The study product is contained in capsules. Each capsule contains either placebo or 40 mg Debio 1450. After fasting overnight, the first two participants in the group receive their capsules. One gets Debio 1450 and one gets Placebo. If these participants tolerate side effects for 24 hours, the remaining six participants receive their assigned capsules.

The plan is to increase the dose for the next group. The study doctor reviews the measurements collected from each group after three days. He may decide to repeat, increase, or lower the dose or even stop the study. The most any participant receives is 800 mg in 20 capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult
2. Has met protocol-specified criteria for qualification and use of contraception
3. Is willing and able to remain confined in the study unit for the entire duration of the treatment period and comply with restrictions related to food, drink and medications
4. Has voluntarily consented to participate and provided written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

1. Has screening laboratory values outside protocol-specified limits
2. Has history of a clinically significant allergic drug reaction
3. Has donated a volume of plasma or whole blood within a time frame not allowed per protocol
4. Has historical or current use not allowed per protocol of:

   1. over-the-counter medications
   2. certain foods; dietary, mineral or herbal supplements
   3. licit or illicit drugs (including experimental drugs, caffeine, nicotine and alcohol)
5. Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

   1. the safety or well-being of the participant or study staff
   2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
   3. the analysis of results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with at least one treatment emergent adverse event (TEAE) | within 10 days post-dose
Maximum observed plasma concentration (Cmax) of Debio 1450 | within 60 hours post-dose
Time of maximum observed plasma concentration (tmax) of Debio 1450 | within 60 hours post-dose

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
  Categorical results will include from time zero to 24 hours post-dose (AUC0-24), from time zero to the last measured concentration (AUC0-t), and from time zero extrapolated to infinity (AUC0-∞).
Percentage of AUC0-∞ that is due to extrapolation beyond the last quantifiable concentration measurement (%AUCex) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Elimination half-life (t½) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Terminal elimination rate constant (λz) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Mean residence time (MRT) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Apparent clearance following oral administration (CL/F) of Debio 1450 | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Apparent volume of distribution of Debio 1450 during terminal phase (Vz/F) | pre-dose, 15, 30 and 60 minutes post-dose, and 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48 and 60 hours post-dose
Cumulative amount of unchanged Debio 1450 excreted in urine (Ae) | pre-dose and 0-2, 2-6, 6-12, 12-24, 24-48 and 48-60 hours post-dose
Percentage of cumulative amount of unchanged Debio 1450 excreted in urine (Ae%) | pre-dose and 0-2, 2-6, 6-12, 12-24, 24-48 and 48-60 hours post-dose
Renal clearance following oral administration | pre-dose and 0-2, 2-6, 6-12, 12-24, 24-48 and 48-60 hours post-dose
Number of participants with clinically significant change from baseline in vital signs | within 10 days post-dose
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) parameters | within 48 hours post-dose
Number of participants with clinically significant change from baseline in clinical laboratory parameters | within 51 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Azra Hussaini, MD, Principal Investigator — Early Phase Clinical Unit - Baltimore, USA
Locations (1):
- Early Phase Clinical Unit, Baltimore, Maryland, United States